CLINICAL TRIAL: NCT01268462
Title: Use of Heliox Associated With PEEP in Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Armele de Fátima Dornelas de Andrade, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31012010
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-10

CONDITIONS: Asthma; Helium; Oxygen; Positive End-Expiratory Pressure
MeSH Terms: conditions — Asthma | interventions — heliox; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Heliox + PEP (Group 1) (Experimental)
  Interventions: Other: Heliox+PEP
- Oxygen+PEP(Group 2) (Experimental)
  Interventions: Other: Oxygen+PEP
- Heliox ( Group 3) (Experimental)
  Interventions: Other: Heliox
- Oxygen (Group 4) (Active Comparator)
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Heliox+PEP — For the nebulization with heliox was used radioaerosol a noninvasive delivery system that consists of a nontoxic orofacial mask with two unidirectional valves - inspiratory and expiratory branch - connected to the nebulizer for radioisotopes Venticis ® II Medical device, class II, CE 0459 (Ventibox / CIS Bio International, France). This mask was attached to the patient's face to prevent leaks and maintain proper pressurization and better patient compliance to the PEP. PEP was offered to 10 cm H2O through valve (Vital Signs, Totowa, NY) attached to the expiratory branch. The nebulizer was fed by a flow of 11 l / min of heliox for the heliox group according to the protocol of Hess et al. When powered by heliox mixture, the flow was adjusted flowmeter suitable for this mixture.
  Arms: Heliox + PEP (Group 1)
Other: Oxygen+PEP — For nebulization of radioaerosol with oxygen, we used a noninvasive delivery system that consists of a mask with two nontoxic orofacial unidirectional valves - inspiratory and expiratory branch - connected to the nebulizer for radioisotopes Venticis ® II Medical device, class II, CE 0459 (Ventibox / CIS Bio International, France). This mask was attached to the patient's face to prevent leaks and maintain proper pressurization and better patient compliance to PEP (Figure 2). PEP was offered to 10 cm H2O through valve (Vital Signs, Totowa, NY) attached to the expiratory branch. The nebulizer was fed by a stream of 8 l / min oxygen.
  Arms: Oxygen+PEP(Group 2)
Other: Heliox — For the nebulization with heliox we used a noninvasive delivery system that consists of a nontoxic orofacial mask with two unidirectional valves - inspiratory and expiratory branch - connected to the nebulizer for radioisotopes Venticis ® II Medical device, class II, CE 0459 (Ventibox / CIS Bio International, France). We used a PEP valve without resistance.
  Arms: Heliox ( Group 3)
Other: Oxygen — For nebulization of radioaerosol with oxygen, we used a noninvasive delivery system that consists of a mask with two nontoxic orofacial unidirectional valves - inspiratory and expiratory branch - connected to the nebulizer for radioisotopes Venticis ® II Medical device, class II, CE 0459 (Ventibox / CIS Bio International, France). We used a PEP valve without resistance.
  Arms: Oxygen (Group 4)

SUMMARY:
In patients with obstructive lung disease like asthma aerosol therapy is the most used for drug administration. A order to make better use of aerosolized drugs in asthmatic patients, studies focus on ways to optimize this administration. Objective: To evaluate the efficacy of nebulized bronchodilators carried by heliox associated with positive expiratory pressure (PEP) in lung deposition of radiation activity in adult asthmatic patients between episodes and its impact on lung function. Methods: A randomized controlled trial involving 32 with a mean age of 47.28 ± 9.67 of which 25% of the sample are male, these patients were divided into four groups: heliox + PEP, + PEP oxygen, heliox and oxygen in Regarding the anthropometric characteristics, parameters and cardiopulmonary baseline spirometry data were similar for all groups. For inhalation lung scintigraphy was used a noninvasive delivery system - orofacial mask with two unidirectional valves nontoxic - inspiratory and expiratory branch - connected to the nebulizer for radioisotopes associated with PEP of 10 cm H2O. At the end of inhalation, the images were acquired in a scintillation camera at 0, 15, 30, 45 and 60 min. In order to analyze the aerosol deposition in different lung areas were delineated regions of interest (ROIs) in the vertical - the upper, middle and bottom - and horizontal central, intermediate and peripheral. Results: The spirometric data showed an increase in the values of forced expiratory volume in one second (FEV1) predicted when compared with the heliox group + PEP (80%, p = 0.030) with PEP + O2 (65%, p = 0.030). As for CI, there was also an increase in PEP + heliox group (0.05 L, p = 0.012) compared to groups without oxygen and heliox PEP (0.03 L, 0.03 L, p = 0.012 respectively) for the total number of counts, no differences were seen between groups with heliox and oxygen with PEP PEP (482510, 577598, p = 0.262 respectively) for the total number of counts by comparing the oxygen group + PEP (577,598) with the heliox group (332,951, p = 0.004) and oxygen without PEP (409,526, p = 0.045), there was a greater number of counts in the O2 + PEP group. By analyzing the rate of pulmonary deposition (IDP) in the vertical gradient, higher deposition in the middle third (p = 0.001) when compared to upper and lower in both groups. With regard to IDPs in the horizontal gradient, there was greater deposition in the intermediate region when compared to central and peripheral (p = 0.003, 0.001 respectively) in all groups. As the penetration rate, no significant differences between groups (p = 0.726). When considering the pulmonary clearance, decreased with the number of counts over time within groups (p <0.05) but no differences between them: heliox + PEP (20.67%), PEP + oxygen (13.50%), heliox (16.27%) and oxygen (16%) - (p> 0.05). Conclusion: Although no differences in the rate of penetration and clearance of pulmonary radiation activity between groups, we noted a higher number of counts in patients who underwent nebulization with oxygen associated with PEP and a functional improvement in patients who underwent nebulization with PEP as spirometric values and CI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of persistent asthma
* FEV1 <60% predicted more than one year
* Reversibility of bronchial obstruction after administration of bronchodilators at least 10% in FEV1 on spirometry.

Exclusion Criteria:

* patients unable to understand or perform the spirometric maneuver or failed to keep in proper positioning to obtain the scintigraphic images
* History of smoking over the past three years associated with a consumption greater than 100 cigarettes per year or who had history of smoking increased 10 years
* pulmonary comorbidities such as COPD, bronchiectasis and tuberculosis sequelae
* Pregnancy and any contraindication to the use of PEP, such as active hemoptysis, sinusitis, surgery or facial trauma, oral or injury, epistaxis, esophageal surgery and nausea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary deposition radioaerosol | 6 mouths
  For inhalation lung scintigraphy, was administered an average dose of acid dietilnotriaminopentaacético labeled with Technetium (DTPA - 99mTc) from 25 to 10 mCi associated bromide drops and 20 drops of Fenoterol bromide ipatropium diluted to a total of up to 3 ml saline 0.9%.

SECONDARY OUTCOMES:
Pulmonary Function | The patient was the pulmonary function test before and after intervention.
  To obtain spirometric values and CI were asked the patients to perform three maneuvers. Spirometry were analyzed FEV1, PEF and forced vital capacity (FVC), considering the percentage of predicted as the best value recorded in accordance with American Thoracic Society. For CI, this correction was performed by body mass index (BMI) and weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Piva JP, Menna Barreto SS, Zelmanovitz F, Amantea S, Cox P. Heliox versus oxygen for nebulized aerosol therapy in children with lower airway obstruction. Pediatr Crit Care Med. 2002 Jan;3(1):6-10. doi: 10.1097/00130478-200201000-00002. PMID 12793914
- [Result] Hess DR, Acosta FL, Ritz RH, Kacmarek RM, Camargo CA Jr. The effect of heliox on nebulizer function using a beta-agonist bronchodilator. Chest. 1999 Jan;115(1):184-9. doi: 10.1378/chest.115.1.184. PMID 9925082
- [Derived] Alcoforado L, Brandao S, Rattes C, Brandao D, Lima V, Ferreira Lima G, Fink JB, Dornelas de Andrade A. Evaluation of lung function and deposition of aerosolized bronchodilators carried by heliox associated with positive expiratory pressure in stable asthmatics: a randomized clinical trial. Respir Med. 2013 Aug;107(8):1178-85. doi: 10.1016/j.rmed.2013.03.020. Epub 2013 May 9. PMID 23664767
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed